CLINICAL TRIAL: NCT05586412
Title: Evaluation of Auricular Vagus Nerve Stimulation and the Effectiveness of Home Exercise Program in Frozen Shoulder Patients
Brief Title: Efficacy of Auricular Vagus Nerve Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burak Buğday, lecturer, Inonu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021/126
Record Dates: First submitted 2022-08-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Being in the 18-50 Age Population; Being Diagnosed With Frozen Shoulder by a Specialist Physician; Volunteer to Participate in the Study
Keywords: frozen shoulder; valgus nerve stimulation; transcutaneous; auricular; home exercises program
MeSH Terms: conditions — Bursitis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomization will be made by drawing lots. 30 patients will be included in the exercise group, 30 patients in the vagus stimulation group, and 30 patients in the exercise and vagus stimulation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise therapy group (Experimental): Exercise therapy group; joint range of motion exercises including the upper extremity, strengthening, stretching, isometric and posture exercise program will be given. These exercises are in the form of a home program and will be asked to do 2 sets a day, 5 days a week, and 10 repetitions of each movement for 4 weeks.
  Interventions: Device: vagus nerve stimulation
- vagus stimulation group (Experimental): To the patients in the vagus stimulation treatment group; Auricular vagus nerve stimulation in the physical therapy and rehabilitation unit, 20 sessions in total, 5 days a week, and 30 minutes each session. will be applied. Patients will be treated in the form of daily arrival and departure. Vagus nerve stimulation will be performed using a TENS device with specially designed ear-shaped surface electrodes, the size of which can be selected according to any size ear. The electrodes will be placed on the inner and outer surface of the tragus and the concha. Waveform biphasic asymmetrical, pulse duration less than 500 microseconds and frequency of 10 hertz for 30 minutes. been applied continuously throughout and the amplitude will be adjusted according to the sensory threshold level.
  Interventions: Device: vagus nerve stimulation
- exercise-vagus stimulation group (Experimental): Exercise and vagus stimulation treatment group; Both the applications made to the patients in the vagus stimulation group and the same exercises given to the patients in the exercise therapy group will be given as a home program. Patients in all groups will be evaluated with different parameters twice, before and after the treatment.
  Interventions: Device: vagus nerve stimulation

INTERVENTIONS:
Device: vagus nerve stimulation — Vagus stimulation, TENS device with specially designed and shaped surfaces that can be shaped according to the magnifying ear will be performed. The electrodes will be placed in such a way that the tragus is facing the inner and outer world. The wave formula is biphasic asymmetrical, pulses less than 500 microseconds and 10 hertz for 30 minutes. will be custom-made and the amplitude will be set as the sensory threshold.
  Other Names: exercise therapy group; exercise-vagus stimulation group

SUMMARY:
Auricular Vagus Nerve Stimulation, a non-invasive method, will be used in the study. Studies have shown that vagus nerve stimulation combined with a large vagal nerve network can have a neuromodulatory effect that will activate some natural protective pathways to improve health. Clinically, vagus nerve stimulation is FDA-approved for epilepsy, treatment-resistant depression, and morbid obesity. Since OSS dysfunction is also involved in the etiology of DO and there is no study on the effectiveness of vagus nerve stimulation in this disease, this study is planned to reveal the effectiveness of auricular vagus nerve stimulation and home exercise program in DO patients.

DETAILED DESCRIPTION:
The shoulder junction is a very dynamic structure that has a wide arc of motion and can move in sagittal, vertical and transverse planes, and provides the connection between the trunk and the upper extremity. Due to this dynamic structure, the shoulder junction is a joint where soft tissue pathologies are common. One of the most common of these pathologies is adhesive capsulitis or frozen shoulder (DO). DO has been defined by different names and with some minor differences in the literature for over 100 years. It has been defined by various names such as adherent obliterative bursitis, adhesive bursitis, periarticular fibrositis, scapulohumeral periarthritis, Duplay periarthritis, adhesive capsulitis. DO was first defined as "scapulohumeral periarthritis" in 1896 by Duplay. In 1934, Codman used the term "frozen shoulder" and suggested that it is seen together with rotator cuff tendinitis. The most widely accepted is the definition made by Neviaser in 1945. It is a disease picture characterized by pain and limitation of movement in the shoulder joint, which is defined as inflammation in the capsule and synovium first, followed by adhesion formations, especially in the axillary fold and the attachment of the capsule to the anatomical neck of the humerus.

Although the exact mechanism of action of vagus nerve stimulation is not known, studies on humans have shown that it affects many areas of the brain at the subcortical and cortical level. A high peripheral sympathetic tone causes regional ischemia, which causes widespread pain. Therapeutic interventions that result in vasodilation (eg, exercise) and appropriate autonomic changes have proven to be effective on pain. The vagus nerve, the "great perfect protector" of the body, encompasses a complex neuro-endocrine-immune network that maintains homeostasis. With reciprocal neural connections to multiple areas of the brain, the vagus nerve serves as a control center that integrates sensitive information and provides appropriate feedback responses. Recent studies show that the vagus nerve is involved in inflammation, mood and pain regulation. All of these can be modulated with vagus nerve stimulation. Vagus nerve stimulation, together with an extensive vagal nerve network, can exert a neuromodulatory effect that will activate some natural protective pathways for health restoration.

Recent preclinical studies show that vagus nerve stimulation is very potent and effective in modulating pain in humans. A medical device allowed the auricular branch of the vagus nerve to be stimulated without any surgery. As a result, it was found that the pain threshold increased and the mechanical pain sensitivity decreased. As a result of the studies, there is a possibility that Frozen Shoulder is a disease that occurs with OSS disorder. Vagus nerve stimulation can be used as an adjunct therapy to correct OSS disorder. Since there is no study in the literature on vagus nerve stimulation in Frozen Shoulder, such a study was considered.

ELIGIBILITY:
Inclusion Criteria:

* To be in the 18-50 age population, to be diagnosed with Frozen Shoulder by a specialist physician

Exclusion Criteria:

* Patients with neurological deficits, neuropathic disorders, chronic inflammation, other musculoskeletal disorders in the upper extremities, pregnant women, and patients who had additional changes in their current treatment other than vagus nerve stimulation were excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-11-03 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
kinesiophobia assessment | 6 months
  Tampa Kinesiophobia Scale were used. The Tampa Kinesiophobia Scale (TKS) is one of them, and it's commonly used in the literature to assess kinesiophobia. It has 17 questions designed to assess fear of moving.
Pain Assessment | 6 months
  Pain Assessment Visual Analogue Scale (VAS) was used. On a 10-centimeter (cm) horizontal line, start 0 (no pain) and finish 10 (unbearable pain) are marked and the subjects were asked to place a mark on this horizontal line according to the degree of pain they felt. The point marked on the line was then measured with the help of a ruler and recorded as the VAS value in cm.
Depression Assessment | 6 months
  Depression Severity Assessment, The Beck Depression Inventory (BDI) was employed, which consists of 21 questions. The scale has a range of 0 to 84 points.
joint range of motion assessment | 6 months
  ROM will be evaluated with the goniometric measurement. This measurement method is an objective method used in the clinical evaluation of joint range of motion. Shoulder flexion, extension, abduction, adduction, external and internal rotation movements of the patients will be measured 3 times passively and actively with a universal goniometer.
functional limitation and disability status assessment | 6 months
  In our study, the Arm, Shoulder and Hand Problems Questionnaire (DASH), which is more preferred in the clinic, was used to evaluate upper extremity functional limitation and disability, which consists of 3 parts. The questionnaire consists of 30 questions that determine the function score in the first part; 21 questions about difficulty in activities of daily living, 5 questions about symptoms (pain, tingling, stiffness, activity-related pain), each of the remaining questions evaluates the patient's social function, work, sleep and self-confidence. The second part of the questionnaire is answered optionally and is a business model consisting of 4 questions. In the third part of the questionnaire, there is a section consisting of 4 elective questions that determine the disability level of patients who are sports-musician models, who want high performance, who are involved in sports or music.
Quality of Life assessment | 6 months
  In our study, the widely preferred SF-36 form, consisting of 36 items, was used to evaluate the quality of life in patients with musculoskeletal disorders, whose reliability and validity have been demonstrated by studies. The 36 items in this form cover 8 different health-related dimensions: physical, emotional and social function, physical role, mental health, general health, pain and vitality. For these dimensions, the scores of the items are coded and converted into a scale between 0-100 points. The scale that evaluates the scores of each subgroup between 0-100; 0 indicates "worst health" status, 100 indicates "best health" status.
Shoulder Pain and Disability Assessment | 6 months
  The Shoulder Pain and Disability Index, developed by Roach et al. in 1911, was used to assess the level of disability by questioning the level of limitation experienced by the participants during personal carrying, care and dressing activities, and to measure current shoulder pain and disability. The Spadi scale consists of 2 subscales of pain (5 questions) and disability (8 questions) and 13 subheadings. Pain and disability subscales are calculated between 0 (no pain) - 100 (worst pain imaginable). As a result of the survey, 3 different scores are obtained as Obstacle, Pain and Total score, each of which is scored separately. The answers given to the questions in the scale are calculated as the last percentile. The higher the total score on the scale, the higher the person's level of pain or disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Malatya Sevgi Hospital, Malatya, Battalgazi̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No